CLINICAL TRIAL: NCT05065567
Title: A Comparison of Haloperidol 5mg IM vs Droperidol 2.5mg and Ondansetron for the Treatment of Hyperemesis in Cannabis Hyperemesis Syndrome
Brief Title: Haloperidol, Droperidol, Ondansetron in Cannabis Hyperemesis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lost too many patients to follow up, unable to enroll enough patients
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EGME#02-2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cyclic Vomiting Syndrome
MeSH Terms: conditions — Familial cyclic vomiting syndrome | interventions — Droperidol; Haloperidol; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- haloperidol (Active Comparator): these patients will receive 5mg IM haloperidol
  Interventions: Drug: Haloperidol
- droperidol (Active Comparator): these patients will receive 2.5mg IV droperidol
  Interventions: Drug: Droperidol
- ondansetron (Active Comparator): these patients will receive 8mg IV ondansetron
  Interventions: Drug: Ondansetron 8mg

INTERVENTIONS:
Drug: Droperidol — Patients with suspected cannabis hyperemesis syndrome and enrolled in the study will be randomized based on the week to 2.5mg droperidol IV
  Arms: droperidol
Drug: Haloperidol — Patients with suspected cannabis hyperemesis syndrome and enrolled in the study will be randomized based on the week to 5mg haloperidol IM
  Arms: haloperidol
Drug: Ondansetron 8mg — Patients with suspected cannabis hyperemesis syndrome and enrolled in the study will be randomized based on the week to ondansetron
  Arms: ondansetron

SUMMARY:
The purpose of this study is to compare two commonly used agents for the treatment of cyclic vomiting to see if one agent is inferior to the other in time to improvement in symptoms, need for repeat or rescue medications, treatment failures and complications/side effects.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with clinical diagnosis of cyclic vomiting in the ED

Exclusion Criteria:

* pregnancy, allergy to any of the study medicines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Haloperidol | Droperidol | Ondansetron
Started | 11 | 14 | 7
Completed | 1 | 5 | 1
Not Completed | 10 | 9 | 6
Not completed — Lost to Follow-up | 10 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol | Droperidol | Ondansetron | Total
Number analyzed (Participants) | 11 | 14 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.45 (8.56) | 29.93 (9.52) | 27.57 (9.52) | 30.28 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 5 | 16
  Male | 9 | 5 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 3 | 15
  White | 5 | 6 | 4 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 7 | 32
Pain_Before_Medication [Mean (Standard Deviation); unit: units on a scale: 0 through 10] | 4.00 (3.30) | 3.38 (3.04) | 4.80 (3.70) | 3.86 (3.17)
Nausea_Before_Medication [Mean (Standard Deviation); unit: units on a scale: 0 through 10] | 3.4 (3.37) | 3.69 (2.50) | 5.00 (4.10) | 3.86 (3.11)

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Pain
Description: change in abdominal pain on 0 (no pain) through 10 (worse possible pain) on a visual analog scale
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 10 | 13 | 5
score on a scale | 4.00 (3.30) | 3.38 (3.04) | 4.8 (3.70)

2. Primary Outcome: Nausea
Description: change in nausea on 0 (none) through 10 (worse possible nausea) on a scale
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 10 | 13 | 6
score on a scale | 3.40 (3.37) | 3.69 (2.50) | 5 (4.10)

3. Secondary Outcome: Treatment Success
Description: both abdominal pain and nausea scores under 2 (none or minimal)
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 11 | 14 | 7
Participants | 2 | 3 | 1

4. Primary Outcome: Abdominal Pain
Description: change in abdominal pain on 0 (no pain) through 10 (worse possible pain) on a visual analog scale
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 1 | 5 | 1
score on a scale | 5 (NA) — Only 1 pt; cannot calculate SD | 2.6 (3.71) | 3 (NA) — Only 1 pt; cannot calculate SD

5. Primary Outcome: Nausea
Description: change in nausea on 0 (none) through 10 (worse possible nausea) on a scale
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 1 | 5 | 1
score on a scale | 3.0 (NA) — Only 1 pt; cannot calculate SD | 3.0 (3.67) | 7.0 (NA) — Only 1 pt; cannot calculate SD

6. Primary Outcome: Abdominal Pain
Description: change in abdominal pain on 0 (no pain) through 10 (worse possible pain) on a visual analog scale
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 1 | 5 | 1
score on a scale | 0 (NA) — Only 1 pt; cannot calculate SD | 3.69 (4.10) | 2 (NA) — Only 1 pt; cannot calculate SD

7. Primary Outcome: Nausea
Description: change in nausea on 0 (none) through 10 (worse possible nausea) on a scale
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 1 | 5 | 1
score on a scale | 0.5 (NA) — Only 1 pt; cannot calculate SD | 3.2 (3.42) | 1 (NA) — Only 1 pt; cannot calculate SD

8. Secondary Outcome: Treatment Success
Description: both abdominal pain and nausea scores under 2 (none or minimal)
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 1 | 5 | 1
Participants | 0 | 3 | 0

9. Secondary Outcome: Treatment Success
Description: both abdominal pain and nausea scores under 2 (none or minimal)
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Droperidol | Ondansetron
Number analyzed (Participants) | 1 | 5 | 1
Participants | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: 48 hours from drug administration.
Arm/Group | Haloperidol | Droperidol | Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/14 | 0/7

LIMITATIONS AND CAVEATS:
Limitations: This study was terminated as the researchers were unable to enroll enough patients and too many patients were lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT05065567/Prot_SAP_002.pdf